CLINICAL TRIAL: NCT05079022
Title: Circulating Tumor DNA (ctDNA)-Minimal Residual Disease (MRD) Based Adjuvant Targeted Therapy in EGFR Mutation-positive Stage I Lung Adenocarcinoma Patients After Complete Surgical Resection
Brief Title: ctDNA-MRD Based Adjuvant Targeted Therapy for EGFR Positive Stage I Lung Adenocarcinomas
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing CSCO-Allist Cancer Research Foundation (Unknown); Shanghai Allist Pharmaceutical Technology Co., Ltd. (Unknown); Guangzhou Burning Rock Medical Examination Institute Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yangfan, Professor of Thoracic Surgery, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Y-2021 AST/zd-0105
Record Dates: First submitted 2021-09-09; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Adenocarcinoma of Lung
Keywords: lung adenocarcinoma; circulating tumor DNA; minimal residual disease; EGFR; furmonertinib
MeSH Terms: conditions — Adenocarcinoma of Lung; Neoplasm, Residual | interventions — aflutinib; AST5902

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Furmonertinib (Experimental): ctDNA-MRD positive participants received 3 years of furmonertinib once daily as adjuvant therapy after radical surgery until disease progression or unacceptable toxicity occurs.
  Interventions: Drug: Furmonertinib

INTERVENTIONS:
Drug: Furmonertinib — Furmonertinib at 80mg dose will be administered orally once daily.
  Other Names: AST2818; AST5902

SUMMARY:
The purpose of this study is to determine the feasibility and effectiveness of ctDNA-MRD based adjuvant furmonertinib therapy in EGFR mutation-positive stage I lung adenocarcinoma patients after complete surgical resection.

DETAILED DESCRIPTION:
Despite surgery provides the best chance for the cure of early-stage lung cancer patients, 20%-40% of stage I non-small cell lung cancer (NSCLC) patients still suffer from disease relapse after R0 resection. One of the important strategies to improve survival is adjuvant therapy.

The adjuvant chemotherapies are reported to improve outcomes of patients with stage II and III lung cancer. However, for stage IA patients, adjuvant chemotherapy is not recommended, while its application in stage IB patients is still controversial. The adjuvant targeted therapy has shown promising effectiveness which can lead to better RFS of EGFR mutation-positive stage IB-IIIA NSCLC patients than chemotherapy in according to several phase III studies. According to the ADAURA study, stage IB NSCLC patients can benefit from the third-generation EGFR-TKI. However, no available study has evaluated the effectiveness of adjuvant targeted therapy in the overall cohort of stage I patients.

Molecular residual disease or minimal residual disease (MRD) refers to residual tumor cells or relative biomarkers that persist in the body after treatment and is below the conventional detection limit. Several studies have confirmed that positive MRD was associated with a poor prognosis. The use of circulating tumor DNA (ctDNA) to reflect MRD at the molecular level can overcome the shortcomings of conventional tests or radiological tests in the detection of recurrence. ctDNA has been proven to detect MRD effectively in stage I-III lung cancer patients and identifying MRD after surgery could facilitate the selection of patients for customized adjuvant therapies.

Thus, the investigators innovatively propose this study to assess the effectiveness of adjuvant targeted therapy (furmonertinib, one third-generation EGFR-TKI) in stage I lung adenocarcinoma patients and explore the role of ctDNA as an MRD monitoring marker in guiding personalized adjuvant therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Stage I lung adenocarcinoma patients underwent complete surgical resection with negative margins (R0) and harbor sensitizing EGFR mutations (exon 19 and/or exon 21).
2. Positive ctDNA after surgery and prior to adjuvant therapy (4 weeks after surgery).
3. Completely recovered from surgery before adjuvant treatment and showed no signs of tumor recurrence in imaging.
4. Adequate organ function: 1) Hemoglobin ≥ 9.0 g/dL; 2)Absolute neutrophil count (ANC) ≥ 1500 cells/mm3; 3) Platelets ≥ 90,000/mm3; 4) AST, ALT ≤ 2.5 x ULN; 5) Total bilirubin ≤ 1.5 x ULN; 6) Serum creatinine ≤ 1.5x ULN and calculated creatinine clearance ≥ 60ml/min.
5. Age >18 years old.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
7. Females must have a negative pregnancy test within 7 days prior to the start of dosing if of child-bearing potential.
8. Males and females of reproductive potential who are sexually active must agree to use adequate contraception prior to entry, during the process and 8 weeks after drug withdrawal.
9. Written informed consent.
10. Compliance with the protocol.
11. Ability to swallow the formulated product.

Exclusion Criteria:

1. Any type of systemic anticancer therapy for lung adenocarcinomas, including chemotherapy, targeted therapy or immunotherapy.
2. Any prior local radiotherapy for lung adenocarcinomas.
3. Clinical objective evidence (pathology or imaging) to confirm disease recurrence before the start of adjuvant therapy.
4. Allergy to furmonertinib or any ingredients.
5. Past medical history of ILD, drug-induced ILD or any evidence of clinically active ILD; CT scan at baseline revealed the presence of idiopathic pulmonary fibrosis.
6. Any evidence of uncontrolled systemic diseases, including active infection, uncontrolled hypertension, unstable angina, angina within the last 3 months, congestive heart failure (≥ New York Heart Association [NYHA] Grade II), myocardial infarction (6 months before enrollment), severe arrhythmia requiring medical treatment, liver diseases, kidney diseases or metabolic diseases.
7. Known history of human immunodeficiency virus (HIV) infection.
8. Pregnant or lactating women.
9. History of neurological or psychiatric disorders, including epilepsy or dementia.
10. Other judgments by the Investigator that the patient should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Clearance of ctDNA at 6 months | 6 months
  To estimate the percentage of patients with undetectable ctDNA at 6 months after adjuvant furmonertinib therapy in stage I lung adenocarcinoma patients who underwent R0 resection and have postoperatively detectable ctDNA prior to adjuvant therapy.

SECONDARY OUTCOMES:
Relapse-free survival (RFS) | Through study completion, an average of 3 years
  To estimate RFS in all postoperative ctDNA-positive stage I lung adenocarcinoma patients, who underwent adjuvant furmonertinib therapy; To compare the RFS in postoperative ctDNA(+) patients who received adjuvant furmonertinib with that in postoperative ctDNA(-) patients, and with that in postoperative ctDNA(+) patients who didn't receive any adjuvant therapy, including chemotherapy, radiotherapy, targeted therapy or immunotherapy.
Clearance of ctDNA at 12 months | 12 months
  To estimate the percentage of patients with undetectable ctDNA at 12 monthsafter adjuvant furmonertinib therapy in stage I lung adenocarcinoma patients who underwent R0 resection and have postoperatively detectable ctDNA prior to adjuvant therapy.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Through study completion, an average of 3 years
  All patients who have received at least one dose furmonertinib will be regarded as the effective population for the safety analysis. Adverse events will be reported and graded in accordance with the NCI common adverse event terminology standard CTCAE version 5.0.
Genomic changes of ctDNA | 0, 3, 6, 12, 18, 24, 30, 36 months
  To dynamically evaluate the ctDNA profiles by next-generation sequencing and illustrate the genomic changes of ctDNA at baseline, during treatment, and at disease relapse.
Relationship between radiomics features and ctDNA status | pre-surgery and 3 days after the surgery
  To evaluate if the radiomics signatures on preoperative CT scans can be a prediction tool for the postoperative ctDNA-MRD status.
Relationship between radiomics features and clinical outcome | pre-surgery and through study completion (an average of 3 years)
  To evaluate if the radiomics signatures on preoperative CT scans can be a prediction tool for relapse-free survival of stage I lung adenocarcinoma patients with R0 resection.

CONTACTS AND LOCATIONS:
Overall Officials: Fan Yang, MD, Study Director — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China